CLINICAL TRIAL: NCT00965861
Title: SCRI Tissue Testing Registry
Status: Terminated | Type: Observational
Why Stopped: Replaced by a study with a similar design.
Sponsor: SCRI Development Innovations, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: SCRI MISC 39
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Melanoma; Myelodysplastic Syndrome; Multiple Myeloma; Lymphoma
Keywords: Tissue Registry; Tissue Collection; Unknown Primary; Breast; Lung; Gastrointestinal; Bone Marrow Transplant; Chronic Lymphocytic Leukemia; Central Nervous System; Head and Neck; Melanoma; Myelodysplastic syndrome; Multiple Myeloma; Lymphoma; Gynecologic; Genitourinary; Refractory Malignancy
MeSH Terms: conditions — Melanoma; Myelodysplastic Syndromes; Multiple Myeloma; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Potential retention of tissue blocks for future study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: The SCRI Oncology Research Consortium will collect written consent from patients allowing the use of their tumor tissue sample(s) for testing/analysis at a future date.
  Interventions: Other: Tissue Registry Study

INTERVENTIONS:
Other: Tissue Registry Study — If a patient consents to allowing the use of their tumor tissue sample(s) for testing/analysis at a future date, their name and information will be stored electronically in a registry that will be managed by SCRI. SCRI may then use the information contained in this registry (such as disease indication, demographic information, etc.) at any time in the future to select tissue samples on which to perform testing/analyses.

SUMMARY:
Sarah Cannon Research Institute (SCRI) is committed to improvement and excellence in clinical research and correlative science. To this end, the SCRI Oncology Research Consortium will collect written consent from patients allowing the use of their tumor tissue sample(s) for testing/analysis at a future date. Future testing may include assays for newly identified markers of potential prognostic and/or therapeutic value. These markers may be specific to an individual cancer type, or they may be present more generally in cancer and/or other conditions.

DETAILED DESCRIPTION:
Sarah Cannon Research Institute (SCRI) is committed to improvement and excellence in clinical research and correlative science. To this end, the SCRI Oncology Research Consortium will collect written consent from patients allowing the use of their tumor tissue sample(s) for testing/analysis at a future date. Future testing may include assays for newly identified markers of potential prognostic and/or therapeutic value. These markers may be specific to an individual cancer type, or they may be present more generally in cancer and/or other conditions.

This study will consist of a registry of patients who have agreed to allow their tissue sample(s) (even those taken prior to their participation in an SCRI-sponsored trial) to be used by the SCRI Oncology Research Consortium at some point in the future for testing and analysis of expression analysis and/or analysis of tumor markers. The registry will be contained in an electronic database, and will be sorted by disease indication. (Note: Patients will not be asked to return at a future date and have tissue samples collected; rather, SCRI will have the authorization to obtain pre-existing samples).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >= 18 years of age.
* Patients must be able to provide written informed consent.

Exclusion Criteria:

* Not Applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The SCRI Oncology Research Consortium will collect written consent from patients allowing the use of their tumor tissue sample(s) for testing/analysis at a future date.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To establish an electronic registry to store information from patients who have provided their consent allowing use of their tissue sample(s) for future testing. | 120 months
To perform testing on the tissue samples to learn more about specific types of cancer and/or other diseases | 120 months

CONTACTS AND LOCATIONS:
Overall Officials: Howard Burris, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States